CLINICAL TRIAL: NCT00410748
Title: Safety and Tolerability of Long-term Administration of Dilaudid CR (Hydromorphone HCI)
Brief Title: Safety and Tolerability of Long-Term Administration of Hydromorphone HCI CR (Controlled Release)
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Alza Corporation, DE, USA (Industry)
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: CR011623
Record Dates: First submitted 2006-12-12; First posted 2006-12-13 (Estimated); Last update posted 2010-04-27 (Estimated); Status verified 2010-04

CONDITIONS: Pain; Analgesics, Opioid
Keywords: Chronic cancer pain; chronic pain
MeSH Terms: conditions — Pain; Chronic Pain

INTERVENTIONS:
Drug: OROS hydromorphone HCI CR

SUMMARY:
The purpose of study was to characterize the safety and tolerability of long-term repeated dosing of OROS hydromorphone controlled release tablets (8,16,32, and 64 mg) in patients with chronic cancer pain or chronic non-malignant pain.

DETAILED DESCRIPTION:
This was a Phase 3, multicenter, open-label, extension study to characterize the safety and tolerability of long-term, repeated dosing of OROS hydromorphone in patients with chronic cancer or chronic non-malignant pain. Patients with chronic cancer or chronic non-malignant pain had completed an OROS hydromorphone short-term study (DO-104, DO-105, DO-119) of approximately 4 weeks duration. During this study, patients continued to receive the dose of OROS hydromorphone that they had been receiving in the short-term study, with dose adjustments as needed to control pain and adverse events. Patients were treated on an outpatient basis. The study was extended from 1 year to up to 2 years in duration. Monthly evaluations of patients treated with OROS hydromorphone for chronic pain were performed to identify adverse events, construct a safety and tolerability profile, and assess efficacy. Dose adjustments were permitted to provide for disease progression, pain control, and adverse events. Quarterly physical examinations were performed to detect significant changes in the underlying condition of patients or changes that may have been associated with long-term opioid therapy. OROS hydromorphone 24 hour controlled release tablets in 8, 16, 32 and 64 mg were ingested orally daily up to 1 year with dose adjustments as needed to control pain and adverse events.

ELIGIBILITY:
Inclusion Criteria:

* Patients who have chronic cancer or chronic non-malignant pain, including pain associated with AIDS, who have successfully completed a OROS hydromorphone HCI (controlled release) short-term study (i.e. Study DO-104, DO-105, or DO-119)
* Patients who require at least 8 mg of hydromorphone HCI every 24 hours for the management of chronic cancer or chronic non-malignant pain
* Patients whose opioid requirements have been stable as demonstrated in a OROS hydromorphone HCI (controlled release) short-term study

Exclusion Criteria:

* Patients intolerant of or hypersensitive to hydromorphone (or other opioid agonists)
* Patients who are pregnant or breast-feeding
* Patients with any gastrointestinal disorder, including pre-existing severe GI narrowing (pathologic or iatrogenic) that may affect the absorption or transit of orally administered drugs
* Patients with clinically significant impaired renal or hepatic function, Addison's disease, hypothyroidism, prostatic hypertrophy, or urethral stricture
* Patients with any significant CNS disorder, including but not limited to head injury, intracranial lesion, increased intracranial pressure, seizure disorder, stroke within the past 6 months, and disorders of cognition
* Patients who are known active drug abusers or alcoholics

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 388 (Actual)
Dates: Study Completion 2000-06 (Actual)

PRIMARY OUTCOMES:
Effectiveness of OROS hydromorphone was maintained throughout the study. OROS hydromorphone provided moderate pain relief in patients with chronic cancer/chronic non-malignant pain.

SECONDARY OUTCOMES:
Long term administration of OROS hydromorphone was safe and well tolerated.

CONTACTS AND LOCATIONS:
Overall Officials: Alza Corporation Clinical Trial, Study Director — ALZA

REFERENCES:
- [Derived] Wallace M, Moulin DE, Rauck RL, Khanna S, Tudor IC, Skowronski R, Thipphawong J. Long-term safety, tolerability, and efficacy of OROS hydromorphone in patients with chronic pain. J Opioid Manag. 2009 Mar-Apr;5(2):97-105. doi: 10.5055/jom.2009.0011. PMID 19507806